CLINICAL TRIAL: NCT05981989
Title: Epidural Electrical Stimulation for Stroke Patients - Improve Motor and Sensory Function and Alleviate Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Buddhist Tzu Chi General Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB112-125-A
Record Dates: First submitted 2023-08-01; First posted 2023-08-08 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Epidural electrical stimulation (EES) (Experimental): Subjects will be implanted with 16-electrode epidural array in the C6-T1 area of the spinal cord. After surgery, subjects will undergo a structured program of physical rehabilitation and electrical stimulation.
  Interventions: Device: Epidural electrical stimulation (EES)

INTERVENTIONS:
Device: Epidural electrical stimulation (EES) — Subjects will undergo a surgical procedure to implant a system that provides epidural electrical stimulation (EES) of the cervical spinal cord. After surgery, subjects will undergo a structured physical rehabilitation program and electrical stimulation.

SUMMARY:
This study aims to verify whether epidural electrical stimulation (EES) of the cervical spinal cord can activate muscles of the upper limbs in people with hemiplegia following a stroke.

DETAILED DESCRIPTION:
The purpose of this study is to verify whether epidural electrical stimulation (EES) of the cervical spinal cord can activate muscles of the arm and hand in people with hemiplegia following stroke. Participants will undergo a surgical procedure to implant a system that provides epidural electrical stimulation (EES) of the cervical spinal cord. After surgery, Participants will undergo a structured physical rehabilitation program and electrical stimulation. Researchers will quantify the motor potentials in the arm and hand muscles generated by EES of the cervical spinal cord, tune optimal stimulation parameters to induced arm and hand movement, and assess participant motor function of the upper limb with standard clinical tests and simple motor tasks.

ELIGIBILITY:
Inclusion Criteria:

* Between 20 and 70 years of age
* First-ever clinical manifest stroke
* Right or left hemiparesis
* Scores higher than 7 and lower than 45 on the Fugl-Meyer scale.
* Expected will undergo spinal cord stimulation surgery.
* Able to comply with procedures and follow up.
* Stable medical condition without cardiopulmonary disease or dysautonomia that would contraindicate participation in upper extremity rehabilitation or testing activities.

Exclusion Criteria:

* Pregnancy or breast feeding.
* Have Major depressive disorder.
* Had a mental illness within one year or been treated in the past.
* Have significant cognitive impairment (MMSE<24) or serious disease that could affect the ability to participate in study activities.
* Cardiovascular or musculoskeletal disease or injury that would prevent full participation in physical therapy intervention.
* Receiving anticoagulant, anti-spasticity or anti-epileptic medications prior to or throughout the duration of the study.
* Unable to read and/or comprehend the consent form.
* Have concerns about this trial and do not sign consent.
* Presence of joint contractures deemed by study clinician/investigator to be too severe to participate in study activities.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in motor functioning and sensation as measured by the Fugl-Meyer Assessment (FMA) | Time Frame: Baseline; at 1 - 4 - 7 - 13 - 19 - 25 months after the implantation
  The Fugl-Meyer Assessment (FMA) is a stroke-specific, performance-based impairment index. It is main assesses motor functioning and sensation in patients with post-stroke hemiplegia. It is applied clinically and in research to determine disease severity, describe motor recovery, and plan and assess treatment. The upper extremity motor function score ranges from 0 to 66.
Change dexterity of the upper limb as measured by the Action Research Arm Test (ARAT) | Time Frame: Baseline; at 1 - 4 - 7 - 13 - 19 - 25 months after the implantation
  Use the Action Research Arm Test (ARAT) assessment to quantify functional hand and arm dexterity. The score ranges from 0 to 57, with a higher value indicating better function.

SECONDARY OUTCOMES:
Change in Quality of Life (QOL) as measured by the World Health Organization Quality of Life (WHOQOL-BREF) | Baseline; at 1 - 4 - 7 - 13 - 19 - 25 months after implantation
  The WHOQOL-BREF is a self-administered questionnaire comprising 26 questions on the individual's perceptions of their health and well-being over the previous two weeks. Responses to questions are on a 1-5 Likert scale where 1 represents "disagree" or "not at all" and 5 represents "completely agree" or "extremely". , The higher the score, the better the quality of life
Change in spasticity as measured by the Modified Ashworth Scale (MAS) | Time Frame: Baseline; at 1 - 4 - 7 - 13 - 19 - 25 months after the implantation
  Quantify spasticity scores using the Modified Ashworth Scale (MAS) for the shoulder, elbow, and wrist. The muscle tension is divided into 0-4 grades. The lower the score, the closer to normal. The higher the score, the more severe the spasticity.

CONTACTS AND LOCATIONS:
Overall Officials: Sheng-Tzung Tsai, M.D., Ph.D., Principal Investigator — Hualien Tzu Chi General Hospital
Locations (1):
- Buddhist Tzu Chi Medical Foundation Hualien Tzu Chi Hospital, Hualien City, Taiwan